CLINICAL TRIAL: NCT06924138
Title: Investigation of the Effect of Functional Respiratory Muscle Training on Functional Level, Balance and Biochemical Parameters in Elderly Individuals.
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Arel University (Other)
Collaborators: Istinye University (Other)
Responsible Party: Principal Investigator, Recep Enes Çelik, Lecturer, Department of Physiotherapy and Rehabilitation, Faculty of Health Sciences, Istanbul Arel University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: IstinyeU
Record Dates: First submitted 2025-03-21; First posted 2025-04-11 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-03

CONDITIONS: Healthy Elderly Individuals
Keywords: functional respiratory muscle training; balance; elderly; oxidative stress; nitric oxide; lactate
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: This study will employ a single-blind design in which participants will be unaware of their group allocation (intervention or control). The intervention and control groups will receive treatments that are identical in appearance and administration procedure to ensure blinding. Investigators will remain unblinded due to the nature of the intervention, which requires close monitoring. This design is intended to minimize bias in participant-reported outcomes and ensure the validity of the findings.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- control group (Active Comparator)
  Interventions: Other: Standart therapy
- intervention group (Experimental)
  Interventions: Other: Exercise; Other: Standart therapy

INTERVENTIONS:
Other: Exercise — The patients included in the study will be randomly divided into two groups as the study and control groups. Randomization will be provided by a computer-aided program. The patients in the study and control groups will be evaluated at the beginning and after six weeks. Functional Respiratory Muscle Training will be given to the study group with the Powerbreathe Respironics® (UK) device. The initial training intensity will be set at 50% (threshold loading) of the MIP value measured in the patient's first evaluation. The patient will be re-evaluated and the new MIP value will be measured, increasing by 10% every 2 weeks, and the training intensity will be adjusted by calculating the measured MIP value. Patients will be asked to work four days a week until the exercise sets are completed.
  Arms: intervention group
Other: Standart therapy — In the control group, the same balance exercises will be performed and will not be changed for six weeks.

SUMMARY:
The aim of this thesis study is to investigate the effects of functional respiratory muscle training on functional level, balance, postural control and biochemical parameters in elderly individuals.

H0 hypothesis: Functional respiratory muscle training has no effect on functional level, balance, postural control and biochemical parameters in elderly individuals.

H1 hypothesis: Functional respiratory muscle training has an effect on functional level, balance, postural control and biochemical parameters in elderly individuals.

The patients included in the study will be randomly divided into two groups as study and control groups. Randomization will be provided by computer-aided program. The patients in the study and control groups will be evaluated at the beginning and after six weeks.

Functional Respiratory Muscle Training will be given to the study group with the Powerbreathe Respironics® (UK) device. The initial training intensity will be set as 50% (threshold loading) of the MIP value measured in the patient's first evaluation. The patient will be re-evaluated and the new MIP value will be measured, increasing by 10% every 2 weeks, and the training intensity will be adjusted by calculating the measured MIP value. Patients will be asked to work four days a week until the exercise sets are completed.

In the control group, the same balance exercises will be performed and will not be changed for six weeks.

DETAILED DESCRIPTION:
When the current literature is examined, it is seen that the relationship between respiration and balance is also exercise applications performed together with inspiratory muscle training. On the other hand, the investigators also come across the effects of different exercises on different biochemical parameters.

However, there is no literature information regarding the parameters that the investigators will evaluate together with functional respiratory muscle training. In addition, although there is no study examining the relationship between functional respiratory muscle training and biochemical parameters, balance, and functional level, the relationship between functional respiratory muscle training and oxidative stress level as a biophysiological acute response and thus changes in endometrial nitric oxide and lactate levels is a significant research topic in the literature. The fact that our study includes a functional respiratory exercise application increases the importance of the study. For this reason, the investigators think that such a study is needed in the literature.

The investigators also hope to contribute to the literature by examining the relationship between functional respiratory muscle training in the elderly population and functional level, balance, and biochemical parameters in our study.

With the functional respiratory muscle training that the investigators will apply for 60 minutes 4 days a week, the investigators expect to protect and maximize the functional level of the patient and the pulmonary dysfunctions, dyspnea symptoms, loss of function that may develop due to peripheral and respiratory muscle weakness in the participants; and as a result, the investigators expect to increase the quality of life. With the study the investigators have determined, the investigators think that the investigators will create a protective preventive exercise protocol to prevent functional losses seen with aging, and at the same time, the investigators will determine the biological infrastructure of the problems encountered and reveal different systematic connections for this. In this way, the investigators aim to both pioneer new studies to be conducted in the literature and contribute to the society and public health by producing scientific data to be used in treatment by clinicians.

ELIGIBILITY:
Inclusion Criteria:

* Being over 65 years of age.
* No cardiopulmonary problems that prevent exercise
* No orthopedic problems that prevent exercise

Exclusion Criteria:

* Being under 65 years of age.
* Presence of cardiopulmonary problems that prevent exercise
* Presence of orthopedic problems that prevent exercise

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Gender Based: Yes — Male, Female
Enrollment: 40 (Estimated)
Dates: Start 2025-02-25 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
Cardiopulmonary exercise test | Baseline and 6 weeks
  Cardiopulmonary exercise testing (CPET) has become an invaluable tool in healthcare, improving disease diagnosis and the quality, efficacy, assessment and safety of treatment in a range of pathologies. The superior ability of CPET to measure the global exercise response of the respiratory, cardiovascular and skeletal muscle systems simultaneously and cost-effectively has led to its application in a variety of settings, from disease diagnosis to preoperative evaluation. In our study, CPET will be applied to assess functional exercise capacity.
Functional Reach Test | Baseline and 6 weeks
  It is a special test that evaluates dynamic balance. The person stands with their feet parallel to a wall. A measuring rod is attached to the wall at shoulder height. The person is asked to lift their arm so that the shoulder is in 90° flexion. The tester marks the patient's fingertip position on the measuring rod. The person is asked to reach forward. The distance reached without losing balance is recorded. While this distance is 45-50 cm on average in healthy people, this distance is shortened in those with balance problems. In the extended version of this test, the anterior, posterior and both lateral directions are measured.
Functional Reach Test Under Load | Baseline and 6 weeks
  The test is defined as the maximum distance that the individual can reach forward in the horizontal plane while maintaining stability on the support surface in the standing position. The patient stands with the arm flexed at 90 degrees and the fist closed, without touching the wall but close to it. The assessor marks the head of the 3rd metacarpal on the wall and the patient is asked to reach forward as far as he can without taking a step, holding a weight with his hands that will be 5% of his body weight. The assessor marks the head of the third metacarpal on the wall again and the difference between the beginning and the end is measured with a tape measure. Three trials are performed and the average of these trials is taken. These tests have been stated as valid and reliable tests for postural control and stability.
Prone Modified Bridge Test | Baseline and 6 weeks
  The participant lies face down with his hands and feet shoulder width apart. The participant is then asked to raise his body off the ground by rising on his hands, forearms and knees. The stopwatch is started. If there is any deterioration in position, the stopwatch is stopped and the test is terminated. The elapsed time is recorded in seconds.
Flamingo Balance Test | Baseline and 6 weeks
  The person stands upright with their hands at waist level. They are asked to lift one foot and place it on the knee of the other leg. The time it takes to stand on one foot without losing balance with their eyes closed is recorded.
Evaluation of the lumbar multifidus and transversus abdominus muscles | Baseline and 6 weeks
  Assessment of Muscles with Stabilizer:
  The Stabilizer Pressure Biofeedback Unit (PBU) will be used to assess the lumbar multifidus and transversus abdominus muscles. The device consists of a three-chambered, air-filled pressure pad, a thin tube carrying the air, and a pressure gauge indicator. The pressure change in the device is reflected to the indicator by the pressure gauge indicator during position or movement change. The device is placed under the lumbar vertebrae in the supine position with the knees flexed and the manometer pressure is set to 40 mmHg. The participant is asked to hold the pressure at this level by contracting the abdominal wall and the time it takes until the deterioration occurs is recorded in seconds.
MIP Measurement | Baseline and 6 weeks
  The maximum inspiratory muscle strength (MIP) of the individuals will be measured using an intraoral pressure measuring device (Microrpm). Intraoral pressure measurement for MIP values has been reported as a valid and reliable method of assessing respiratory functions within the scope of the American Thoracic Society/European Respiratory Society (ATS/ERS) protocol. During the MIP measurement, the individual is asked to make a maximum expiration and then a maximal inspiration with a nose clip and maintain this for 1-3 seconds.
MEP Measurement | Baseline and 6 weeks
  The maximum expiratory muscle strength (MEP) of the individuals will be measured using an intraoral pressure measuring device (Microrpm). Intraoral pressure measurement for MEP values has been reported as a valid and reliable method of assessing respiratory functions within the scope of the American Thoracic Society/European Respiratory Society (ATS/ERS) protocol. During the MEP measurement, the individual is asked to make a maximum expiration and then a maximal inspiration with a nose clip and maintain this for 1-3 seconds.
Total Antioxidant Capacity | Baseline and 6 weeks
  Inflammation, nutrients, normal metabolism, spreading, aging, high oxygen pressure (pO2), ozone (O3), nitrogen dioxide (NO2), chemical substances, cigarettes and storage of many stimuli such as storage, molecules called oxidants emerge. These oxidant molecules are called free radicals or reactive oxygen species (ROS).
  Oxidants: can damage all important images such as lipid, protein, DNA, resolution and enzyme; they can lead to dozens of important problems such as cancer, heart diseases, shoot diseases, structural disorders in the vessels and premature aging.
Total Oxidant Level | Baseline and 6 weeks
  The oxidants in the sample oxidize the ferrous ion-o-dianisidine complex to ferric ion. The glycerol in the medium accelerates this reaction by approximately three-fold. Ferric ions form a colored complex with xylenol orange in an acidic medium. The intensity of the color, which is related to the amount of oxidants in the sample, is measured spectrophotometrically.
  At the time of the study, the samples previously stored at -80 ºC will be brought to room temperature.
  - 15 µl of the standard and samples will be taken and pipetted into the microplate.
Measurement of Endothelial Nitric Oxide levels | Baseline and 6 weeks
  During the experimental phase, samples will be thawed and lactate and eNOS levels in the samples will be measured by a commercial ELISA-based kit. Briefly; samples and standards will be added to appropriate wells pre-coated with Anti-Human monoclonal antibody before incubation. Then, after biotin is added to all wells and combined with Streptavidin-HRP to form immune complex, the plate will be left for incubation. Uncombined enzyme will be removed by washing processes, then Chromogen Solution A and B will be added sequentially to turn the color of the liquid in the wells blue. At the end of the reaction, the color will be yellow due to the effect of acid. Optical density will be read at 450 nm in a plate reader (Thermo Scientific Microplate Reader, USA).
Measurement of Lactate levels | Baseline and 6 weeks
  During the experimental phase, samples will be thawed and lactate and eNOS levels in the samples will be measured by a commercial ELISA-based kit. Briefly; samples and standards will be added to appropriate wells pre-coated with Anti-Human monoclonal antibody before incubation. Then, after biotin is added to all wells and combined with Streptavidin-HRP to form immune complex, the plate will be left for incubation. Uncombined enzyme will be removed by washing processes, then Chromogen Solution A and B will be added sequentially to turn the color of the liquid in the wells blue. At the end of the reaction, the color will be yellow due to the effect of acid. Optical density will be read at 450 nm in a plate reader (Thermo Scientific Microplate Reader, USA).
Berg Balance Scale | Baseline and 6 weeks
  It has 14 stages including sitting without support, transition from sitting to standing, standing without support, standing with eyes closed, standing with feet together, reaching forward, picking up an object on the floor, turning and looking over the right and left shoulders, turning 360◦, touching the step alternatively, heel/toe, standing on one leg, transitioning from standing to sitting, and transfers. The tester observes the patient during the activity and gives scores between 0 and 4.
Tinetti Balance Performance Evaluation | Baseline and 6 weeks
  It is a screening test used to evaluate balance and walking status. The balance section of the test is scored out of 16 points and the walking section is scored out of 12 points, for a maximum of 28 points. Performance is evaluated during sitting without support, standing up from sitting, coming to sitting from standing, standing without support, standing with eyes closed, turning 360 degrees, and sternal thrust.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Arel University, Istanbul, Zeytinburnu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dimitriadis Z, Kapreli E, Konstantinidou I, Oldham J, Strimpakos N. Test/retest reliability of maximum mouth pressure measurements with the MicroRPM in healthy volunteers. Respir Care. 2011 Jun;56(6):776-82. doi: 10.4187/respcare.00783. Epub 2011 Feb 9. PMID 21310113
- [Background] Ceylan, E. (2014). Kardiyopulmoner egzersiz testleri. Journal of Clinical and Experimental Investigations, 5(3), 504-509.
- [Background] Morales CR, Sanz DR, Reguera MC, Martinez SF, Gonzalez PT, Pascual BM. Proprioceptive Stabilizer training of the abdominal wall muscles in healthy subjects: a quasi-experimental study. Rev Assoc Med Bras (1992). 2018 Dec;64(12):1134-1138. doi: 10.1590/1806-9282.64.12.1134. PMID 30569991
- [Background] Leelarungrayub J, Puntumetakul R, Sriboonreung T, Pothasak Y, Klaphajone J. Preliminary study: comparative effects of lung volume therapy between slow and fast deep-breathing techniques on pulmonary function, respiratory muscle strength, oxidative stress, cytokines, 6-minute walking distance, and quality of life in persons with COPD. Int J Chron Obstruct Pulmon Dis. 2018 Dec 5;13:3909-3921. doi: 10.2147/COPD.S181428. eCollection 2018. PMID 30584292
- [Background] van Helvoort HA, van de Pol MH, Heijdra YF, Dekhuijzen PN. Systemic inflammatory response to exhaustive exercise in patients with chronic obstructive pulmonary disease. Respir Med. 2005 Dec;99(12):1555-67. doi: 10.1016/j.rmed.2005.03.028. PMID 15890510
- [Background] Heidari B. The importance of C-reactive protein and other inflammatory markers in patients with chronic obstructive pulmonary disease. Caspian J Intern Med. 2012 Spring;3(2):428-35. PMID 24358439
- [Background] ben Anes A, Fetoui H, Bchir S, ben Nasr H, Chahdoura H, Chabchoub E, Yacoub S, Garrouch A, Benzarti M, Tabka Z, Chahed K. Increased oxidative stress and altered levels of nitric oxide and peroxynitrite in Tunisian patients with chronic obstructive pulmonary disease: correlation with disease severity and airflow obstruction. Biol Trace Elem Res. 2014 Oct;161(1):20-31. doi: 10.1007/s12011-014-0087-4. Epub 2014 Jul 31. PMID 25074430
- [Background] McConnell AK. The role of inspiratory muscle function and training in the genesis of dyspnoea in asthma and COPD. Prim Care Respir J. 2005 Aug;14(4):186-94. doi: 10.1016/j.pcrj.2005.03.008. Epub 2005 Jun 27. PMID 16701724
- [Background] Archiza B, Andaku DK, Caruso FCR, Bonjorno JC Jr, Oliveira CR, Ricci PA, Amaral ACD, Mattiello SM, Libardi CA, Phillips SA, Arena R, Borghi-Silva A. Effects of inspiratory muscle training in professional women football players: a randomized sham-controlled trial. J Sports Sci. 2018 Apr;36(7):771-780. doi: 10.1080/02640414.2017.1340659. Epub 2017 Jun 16. PMID 28622081
- [Background] Rivara MB, Yeung CK, Robinson-Cohen C, Phillips BR, Ruzinski J, Rock D, Linke L, Shen DD, Ikizler TA, Himmelfarb J. Effect of Coenzyme Q10 on Biomarkers of Oxidative Stress and Cardiac Function in Hemodialysis Patients: The CoQ10 Biomarker Trial. Am J Kidney Dis. 2017 Mar;69(3):389-399. doi: 10.1053/j.ajkd.2016.08.041. Epub 2016 Dec 4. PMID 27927588
- [Background] Eickhoff P, Valipour A, Kiss D, Schreder M, Cekici L, Geyer K, Kohansal R, Burghuber OC. Determinants of systemic vascular function in patients with stable chronic obstructive pulmonary disease. Am J Respir Crit Care Med. 2008 Dec 15;178(12):1211-8. doi: 10.1164/rccm.200709-1412OC. Epub 2008 Oct 3. PMID 18836149
- [Background] Campos NG, Marizeiro DF, Florencio ACL, Silva IC, Meneses GC, Bezerra GF, Martins AMC, Liborio AB. Effects of respiratory muscle training on endothelium and oxidative stress biomarkers in hemodialysis patients: A randomized clinical trial. Respir Med. 2018 Jan;134:103-109. doi: 10.1016/j.rmed.2017.12.005. Epub 2017 Dec 7. PMID 29413495
- [Background] Tong TK, McConnell AK, Lin H, Nie J, Zhang H, Wang J. "Functional" Inspiratory and Core Muscle Training Enhances Running Performance and Economy. J Strength Cond Res. 2016 Oct;30(10):2942-51. doi: 10.1519/JSC.0000000000000656. PMID 25162653
- [Background] Zunner BEM, Wachsmuth NB, Eckstein ML, Scherl L, Schierbauer JR, Haupt S, Stumpf C, Reusch L, Moser O. Myokines and Resistance Training: A Narrative Review. Int J Mol Sci. 2022 Mar 23;23(7):3501. doi: 10.3390/ijms23073501. PMID 35408868
- [Background] Tounsi B, Acheche A, Lelard T, Tabka Z, Trabelsi Y, Ahmaidi S. Effects of specific inspiratory muscle training combined with whole-body endurance training program on balance in COPD patients: Randomized controlled trial. PLoS One. 2021 Sep 23;16(9):e0257595. doi: 10.1371/journal.pone.0257595. eCollection 2021. PMID 34555068
- [Background] Mota S, Guell R, Barreiro E, Solanes I, Ramirez-Sarmiento A, Orozco-Levi M, Casan P, Gea J, Sanchis J. Clinical outcomes of expiratory muscle training in severe COPD patients. Respir Med. 2007 Mar;101(3):516-24. doi: 10.1016/j.rmed.2006.06.024. Epub 2006 Aug 30. PMID 16942867
- [Background] Gosselink R, De Vos J, van den Heuvel SP, Segers J, Decramer M, Kwakkel G. Impact of inspiratory muscle training in patients with COPD: what is the evidence? Eur Respir J. 2011 Feb;37(2):416-25. doi: 10.1183/09031936.00031810. PMID 21282809
- [Background] Akgül, A., Tarakci, E., Arman, N., Büyükkaya, F., Irmak, H. S., & Karaaslan, T. (2018). Yaşlılarda denge, mobilite ve düşmenin değerlendirilmesi. Türkiye Klinikleri. Tip Bilimleri Dergisi, 38(1), 94-98.
- [Background] Janssens L, Brumagne S, McConnell AK, Claeys K, Pijnenburg M, Goossens N, Burtin C, Janssens W, Decramer M, Troosters T. Impaired postural control reduces sit-to-stand-to-sit performance in individuals with chronic obstructive pulmonary disease. PLoS One. 2014 Feb 12;9(2):e88247. doi: 10.1371/journal.pone.0088247. eCollection 2014. PMID 24533072
- [Background] Hodges PW, Heijnen I, Gandevia SC. Postural activity of the diaphragm is reduced in humans when respiratory demand increases. J Physiol. 2001 Dec 15;537(Pt 3):999-1008. doi: 10.1111/j.1469-7793.2001.00999.x. PMID 11744772
- [Background] Sieck GC, Ferreira LF, Reid MB, Mantilla CB. Mechanical properties of respiratory muscles. Compr Physiol. 2013 Oct;3(4):1553-67. doi: 10.1002/cphy.c130003. PMID 24265238